CLINICAL TRIAL: NCT03460977
Title: A PHASE I DOSE ESCALATION AND EXPANDED COHORT STUDY OF PF 06821497 (MEVROMETOSTAT) IN THE TREATMENT OF ADULT PATIENTS WITH RELAPSED/REFRACTORY SMALL CELL LUNG CANCER (SCLC), CASTRATION RESISTANT PROSTATE CANCER (CRPC) AND FOLLICULAR LYMPHOMA (FL)
Brief Title: A Study of Mevrometostat for Treatment of Relapsed/Refractory SCLC, Castration Resistant Prostate Cancer, and Follicular Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C2321001; EZH2 (Other: Alias Study Number); 2023-509179-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2018-02-12; First posted 2018-03-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC); Small Cell Lung Cancer (SCLC); Follicular Lymphoma (FL)
Keywords: EZH2; enhancer of zeste homolog 2; castrate resistant prostate cancer; prostatecancer-study.com; mCRPC; efficacy; safety; pharmacokinetics; pharmacodynamics; dose escalation; dose expansion; open-label; small cell lung cancer; SCLC; follicular lymphoma; FL; relapsed; refractory
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lymphoma, Follicular; Recurrence | interventions — PF06821497; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose Escalation (Part 1A) (Experimental): Participants with SCLC, CRPC and FL will receive mevrometostat at escalating dose levels
  Interventions: Drug: Mervometostat (PF-06821497)
- Dose Escalation (Part 1B) (Experimental): Participants with FL will receive mevrometostat at escalating dose levels
  Interventions: Drug: Mervometostat (PF-06821497)
- Dose Escalation (Part 1C) (Experimental): Participants with mCRPC will receive PF-06821497 at escalating dose levels.
  Interventions: Drug: Mervometostat (PF-06821497)
- Dose Escalation (Part 2A) (Experimental): Participants with mCRPC and SCLC will receive mevrometostat at escalating dose levels in combination with SOC.
  Interventions: Drug: Mervometostat (PF-06821497); Drug: Enzalutamide
- Dose Expansion (Part 2B) (Experimental): Participants with CRPC will receive mevrometostat in combination with SOC or SOC alone.
  Interventions: Drug: Mervometostat (PF-06821497); Drug: Enzalutamide
- Japan Cohort (Experimental): Participants with CRPC will receive mevrometostat at one or two doses
  Interventions: Drug: Mervometostat (PF-06821497)
- China cohort (Experimental): Participants will receive mevrometostat at one or two doses
  Interventions: Drug: Mervometostat (PF-06821497)
- Dose Expansion (Part 2C) (Experimental): Participants with mCRPC will receive mevrometostat at a different dose/dosing regimen than that of Part 2B in combination with SOC
  Interventions: Drug: Mervometostat (PF-06821497); Drug: Enzalutamide
- BE Substudy (Experimental): In the assessment phase, each enrolled participant will receive single doses of the 2 different mevrometostat formulations in 3 periods with alternating dosing and washout between each dose. In the maintenance phase, each participant will receive mevrometostat 2 times a day and enzalutamide 1 time a day.
  Interventions: Drug: Mervometostat (PF-06821497); Drug: Enzalutamide
- DDI Substudy (Experimental): In the assessment phase, each enrolled participant will receive a combination of mevrometostat, enzalutamide, and itraconazole based on preset schedule. In the maintenance phase, each participant will receive mevrometostat 2 times a day and enzalutamide 1 time a day.
  Interventions: Drug: Mervometostat (PF-06821497); Drug: Enzalutamide

INTERVENTIONS:
Drug: Mervometostat (PF-06821497) — Oral continuous
  Other Names: EZH2i
Drug: Enzalutamide — Oral continuous
  Other Names: Xtandi
  Arms: BE Substudy; DDI Substudy; Dose Escalation (Part 2A); Dose Expansion (Part 2B); Dose Expansion (Part 2C)

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called Mevrometostat) for the possible treatment of Relapsed/ Refractory Small Cell Lung Cancer (SCLC), Castration Resistant Prostate Cancer (CRPC) and Follicular Lymphoma (FL). The study consists of 3 parts; Part 1 and 2 enrolled participants with SCLC, metastatic CRPC, and FL are closed for enrollment.

Part 3, which is open for enrollment is seeking men who:

* have Castration Resistant Prostate Cancer (CRPC) and
* have previously received treatment for CRPC and have progressed from the last treatment

All participants in Part 3 of this study will receive mevrometostat and/ or enzalutamide. Part 3 consists of 2 sub studies each has an assessment phase and a maintenance phase.

In the assessment phase:

* participants in the BE substudy will take 3 single doses of mevrometostat by mouth over 3 periods.
* participants in the DDI substudy will take mevrometostat 2 times a day, with or without enzalutamide 1 time a day, and/or itraconazole 1 time a day based on a present schedule.

After completion of the assessment phase, participants will enter the maintenance phase where they will receive mevrometostat 2 times a day and enzalutamide 1 time a day by mouth until their cancer is no longer responding.

The studywill look at the experiences of participanrs receiving the study medicine. This will help see if the study medicine is safe and effective.

DETAILED DESCRIPTION:
This is an open label, multi center, Phase 1 dose escalation and dose expansion study of mevrometostat (PF-06821497) administered orally BID as a single agent or in combination with SOC to patients with CRPC, SCLC, and FL. The study consists of three parts (Part 1, Part 2, and Part 3) along with the Japan and China monotherapy cohorts. Part 1 and Part 2 are closed for enrollment. Part 1 tested monotherapy in 3 cohorts (Parts 1A, 1B, and 1C); Part 2 tested combination therapy in Parts 2A (dose escalation), 2B and 2C (does expansion).

Part 3 consists of the Bioequivalence (BE) and drug-drug interaction (DDI) substudies and are open for enrollment. The BE substudy will test between 2 mevrometostat formulation to confirm that they work in the body the same way. The DDI substudy will evaluate the effect of a strong CYP3A4 (an enzyme in your body that breaks down/ removes drugs) inhibitor on the PK of mevrometostat; a strong CYP3A4 inhibitor may slow down the breakdown/ removal of drugs in your body.

ELIGIBILITY:
Part 1 and Part 2 (Closed for enrollment).

Part 3 Key Inclusion Criteria:

* Histological or cytological diagnosis of castration resistant prostate cancer.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2 with expected life expectancy of at least 6 months.
* Adequate bone marrow, renal, and liver function

Part 3 Key Exclusion Criteria:

* Prior irradiation to >25% of the bone marrow.
* QTcF interval >480 msec at screening.
* Hypertension that cannot be controlled by medications (>150/90 mmHg despite optimal medical therapy).
* Known or suspected hypersensitivity to PF 06821497 or any components or enzalutamide (CRPC)
* Active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease or previous gastric resection or lap band surgery.
* Current use or anticipated need for food or drugs that are known strong and moderate CYP3A4/5 inducers or inhibitors
* Prior enzalutamide within the last 4 weeks
* DDI SUBSTUDY:
* history of CHF or evidence of ventricular dysfunction
* fructose intolerance
* coadministration of CYP3A4 substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-03-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with dose limiting toxicities (DLTs) to determine the maximum tolerated dose (MTD) | Baseline up to 90 days
  First cycle DLTs will be utilized to determine the MTD
Overall safety profile including adverse events | Baseline up to approximately 2 years
  Adverse Events will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version [4.03])
Preliminary efficacy determination as evaluated by disease specific response criteria | Through study completion, approximately 2 years past last patient first visit.
  Objective response using Response Evaluation Criteria in Lymphoma (RECIL) for lymphoma, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for solid tumors including Small Cell Lung Cancer (SCLC) and Prostate Cancer Working Group 3 (PCWG3) for Castration Resistant Prostate Cancer (CRPC). Progression-free survival in Part 2B in patients with CRPC.
Overall safety profile including laboratory abnormalities | Baseline up to approximately 2 years
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version [4.03]), and timing.
Overall safety profile including vital signs | Baseline up to approximately 2 years
  Vital sign changes from baseline including blood pressure, heart rate, ECG changes.
Evaluate time to event mevrometostat and enzalutamide vs enzalutamide alone including radiographic prgression free survival | Baseline until disease progression or death or through study completion (approx 2 years)
  PCWG3

SECONDARY OUTCOMES:
Evaluate time to event anti-tumor activity of mevrometostat including progression-free survival (PFS), PSA50, Duration of Response (DoR), Time to first skeletal related event and Time to symptomatic skeletal related event, depending on tumor type. | Baseline and every 21 days through time of confirmed disease progression, unacceptable toxicity, or through study completion, approximately 2 years.
  Time to event endpoints based on Response Evaluation Criteria in Lymphoma (RECIL) for lymphoma, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for solid tumors including Small Cell Lung Cancer (SCLC) and Prostate Cancer Working Group 3 (PCWG3) for Castration Resistant Prostate Cancer (CRPC)
Evaluate overall survival | Baseline up to approximately 2 years
  Median time to death proportion of patients alive at 6 months, 1 year, and 2 years.
Pharmacokinetic Parameters: Maximum Observed Plasma Concentration (Cmax) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Single dose and multiple dose PK will be calculated as data permits
Pharmacokinetic Parameters: Time to Reach Maximum Observed Plasma Concentration (Tmax) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Single dose and multiple dose PK will be calculated as data permits
Pharmacokinetic Parameters: Area Under the Curve (AUC) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Single dose and multiple dose PK will be calculated as data permits
Pharmacokinetic Parameters: Apparent Oral Clearance (CL/F) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Single dose and multiple dose PK will be calculated as data permits
Pharmacokinetic Parameters: Apparent Volume of Distribution (Vz/F) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Single dose and multiple dose PK will be calculated as data permits
Pharmacokinetic Parameters: Plasma Decay Half-Life (t1/2) | At specific timepoints from Cycle 1 day 1 to End of Treatment visit
  Singe dose and multiple dose PK will be calculated as data permits
Evaluate the impact of mevrometostat on patient reported outcomes. | At specific time-points from Cycle 1 Day 1 to End of Treatment visit.
  Quality of Life and Time to Functional Status Deterioration as assessed by FACT-P.
Impact of mevrometostat in combination with enzalutamide, enzalutamide alone and mevrometostat alone on symptoms and symptomatic toxicity | At specific time points from Cycle1 Day 1 to end of treatment
  Questionnaire customized from PRO-CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (44):
  - Banner-University Medical Center Tucson, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Arizona Urology Specialists, PLLC, Tucson, Arizona
  - Pacific Cancer Medical Center INC, Anaheim, California
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - City of Hope Investigational Drug Services (IDS), Duarte, California
  - Norwalk Hospital, Norwalk, Connecticut
  - The University of Kansas Cancer Center, Investigational Drug Services, Fairway, Kansas
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Medical Center Medical Office Building, Kansas City, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute Pharmacy, Downtown Pharmacy, Louisville, Kentucky
  - Norton Cancer Institute Pharmacy, Louisville, Kentucky
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute- Chestnut Hill, Newton, Massachusetts
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - OU Health University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Stephenson Cancer Center (chemo location), Oklahoma City, Oklahoma
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern University Hospital - William P. Clements, Jr, Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Olympic Medical Center, Port Angeles, Washington
  - Fred Hutchinson Cancer Center Alliance Peninsula, Poulsbo, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo, Bulgaria
- China (6):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Poland (4):
  - Szpital Wojewódzki im. Mikołaja Kopernika w Koszalinie, Koszalin
  - Centrum Diagnostyczne Affidea Koszalin, Koszalin
  - Centrum Medyczne MEDYK, Rzeszów
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw
- Russia (9):
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - LLC "Neyro-klinika", Moscow
  - Moscow GBUZ "City clinical hospital n. a. S.P. Botkina" of Moscow health department, Moscow
  - SBHI of Moscow City Clinical Hospital, Moscow
  - Budgetary Healthcare Institution of Omsk region "Clinical Oncological Dispensary", Omsk
  - Federal State Budgetary Institution National Medical Research Center n.a. V.A. Almazov, Saint Petersburg
  - Federal State Budgetary Institution National Medical Research Center for Oncology n.a. N.N., Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City Clinical Oncological Dispensary", Saint Petersburg
  - State Budgetary Healthcare Institution of the Yaroslavl Region, Yaroslavl
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Chungnam national university hospital, Daejeon, Taejǒn-kwangyǒkshi
- Spain (12):
  - Institut Català d´Oncología (ICO)-H. Durán i Reynals, L'Hospitalet de Llobregat, Barecelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hospital Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - H.U. Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321001